CLINICAL TRIAL: NCT02482493
Title: A Prospective Randomised Control Trial to Compare Clinical and Radiological Outcomes of the Press-Fit Condylar All-Polyethylene Tibial Component With Metal-Backed Tibial Component Implant, in Patients Aged 75 Years or Over
Brief Title: All Polyethylene Versus Metal Backed Tibial Components in Knee Replacement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maidstone & Tunbridge Wells NHS Trust (Other)
Responsible Party: Principal Investigator, Helen Samuel, Mr Nick Bowman- Consultant Orthopaedic Surgeon, Maidstone & Tunbridge Wells NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14/01/282 version 1.3
Record Dates: First submitted 2015-06-17; First posted 2015-06-26 (Estimated); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- All-polyethylene Tibial component (Active Comparator): Sigma PFC All polyethylene Tibial component will be implanted
  Interventions: Device: Sigma PFC
- Metal Backed Tibial component (Active Comparator): Sigma PFC metal-backed tibial component will be implanted
  Interventions: Device: Sigma PFC

INTERVENTIONS:
Device: Sigma PFC — patients will receive either an all polyethylene tibial component or a metal- backed component

SUMMARY:
Total knee arthroplasty (TKA) is one of the most commonly performed orthopaedic procedures. Approximately 84,000 knee replacement procedures were recorded in the UK in 2012. The main goal of TKA is to relieve the disabling pain of arthritic disease.

Patient satisfaction following TKA is related to quick recovery and return to daily activities. This can be dependent on the design of the implant used in the knee. Improvements in implant design and surgical technique mean many modern designs offer implant survival rates beyond 10 - 15 years.

As cost pressure increases in the NHS the unit cost of implants is now being scrutinised, particularly with regard to cost effectiveness. The Press-Fit Condylar (PFC) Sigma implant can be used with either a conventional metal backed or alternatively an all polyethylene tibial component (part fitted to the shin bone), the latter considerably cheaper to manufacture. Four small prospective randomised trials and one large regional registry study with long follow up support the safe use of all polyethylene tibial components in TKA. The investigators will therefore undertake a prospective randomised controlled trial comparing the results of all polyethylene tibial components with those of conventional metal backed tibial components in patients aged 75 or over, comparing both clinical outcome and radiological survivorship.

The type of knee replacement used for each patient (metal-backed or polyethylene) will be chosen at random once a patient has agreed to take part in the study.

Data will be collected by means of follow-up appointments and questionnaires and clinical tests both before the operation 1 year, 2 years and 5 years postoperatively. This will allow us to see how both types of knee replacement perform over time and if one performs better than the other in terms of patients movement, pain and functional activities.

DETAILED DESCRIPTION:
Summary of design and methodology.

When a patient who is appropriate for the study is added to the waiting list for a Total Knee replacement they will be given (or if missed, posted) an information sheet about the study. This will allow patients several weeks to read the information and telephone the Orthopaedic research department, if they wish, with any questions they may have.

The Patients will then come to preassessment clinic as usual. At this point the study will be explained again in person, the patient will be given time to ask questions and will be asked if they wish to consent to participating.

If the patient consents to taking part they will complete preoperative measures and questionnaires There are 3 questionnaires on how the patient is functioning. 2 are completed by the patient and 1 with the help of the Researcher

The questionnaires are:

Oxford Knee Score American Knee Society Score (AKSS) Medical Outcomes Study Short Form-36 Health Survey (MOS SF-36) All questionnaires will be performed preoperatively, 1 year, 2 years and 5 years postoperatively.

Six weeks postoperatively the patient will attend a follow-up clinic. This is standard for all patients undergoing knee replacement surgery at the Tunbridge Wells Hospital. Routine wound checks and postoperative care will take place and any patient's concerns dealt with. At this point the patient will be booked in for another routine follow up appointment 3 months postoperatively. No study data will be collected at these visits besides adverse events or lost to follow-up where appropriate.

At one year post-operatively the patient will be asked to attend for an appointment. The knee will be assessed clinical and same series of clinician and patient questionnaires completed. A series of x-rays will also be taken to allow the position of the implant to be recorded. Measurements will be taken to be taken from the x-rays Similarly the patient will be invited to attend a further 2 appointments at 2 year and 5 years post-operatively. At these appointments the questionnaires will be repeated along with the x-rays.

Should the patient wish to withdraw at any point they are free to do so and will not then be contacted for any subsequent appointments unless they are due routine clinical appointments .

Any patient undergoing total knee replacement and not in the study will attend routine 6 week and 3 month and one year follow-up appointments, as routine but will be discharged when appropriate and will not be subject to long term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients suitable for simple cemented primary knee arthroplasty
* Patients presenting with osteoarthritis of the knee
* Patients with inflammatory arthropathy, requiring total knee arthroplasty
* Patients must be ambulatory at time of preoperative assessment clinic
* Patients must be able to understand instructions and be willing to return for follow up
* Patients aged 75 years or over at the time of surgery

Exclusion Criteria:

* Previous knee surgery (except arthroscopic / open meniscectomy)
* Patients with significant medical co-morbidity
* Disorders causing abnormal gait or significant pain
* Patients unable to consent
* Severe visual impairment

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
American Knee Society Score | 5 year outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gibb, Principal Investigator — Maidstone and Tunbridge Wells NHS trust
Locations (1):
- Trauma & Orthopaedic Dept, Tunbridge Wells Hospital, Pembury, Kent, United Kingdom